CLINICAL TRIAL: NCT03798990
Title: Reduce Speed Limits From 90km/h to 80 km/h on French Two-way Roads Without Central Separator: the Number of Traffic Related Fatalities on the Network Concerned "Before and After" the Reduction of Speed Limits.
Brief Title: Reduce Speed Limits From 90km/h to 80 km/h on French Roads: Impact on Mortality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre d'études et d'expertise sur les risques, l'environnement, la mobilité et l'aménagement (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-12
Record Dates: First submitted 2018-12-21; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Health Risks; Death
Keywords: Speed; Road safety
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- users of French roads: all road users circulating on French roads outside over-seas

SUMMARY:
On the first July 2018, the French government lowered the maximum authorized speeds on two-way roads without a central separator from 90 km/h to 80 km/h. The network concerned represents approximately 400 000 km of roads outside the built-up area, accounting for 55% of road deaths.

The objective of the measure is to reduce the number of deaths on the roads concerned by encouraging the reduction of the average speed practiced by drivers.

The analysis deals with a comparison of the number of killed persons on the network concerned, before and after the reduction of the speed limits. The "before" period is 2015-2017. The "after" period is from July 2018 to June 2019.

The data used are extracted from the national bodily injury accident file (BAAC). The police fills this file for each road accidents occurring on a road open to public traffic and causing at least one victim (i.e., one user requiring medical care and involving at least one vehicle).

DETAILED DESCRIPTION:
This measure was intended general and concerns a type of roads in its entirety. The rest of the road network is too heterogeneous (urban, highways ...), leading to an accidentology very far in terms of severity, users concerned and families of accidents to allow the establishment of control groups that would not be affected by a reduction in the speed limit. As a result, the principle of an assessment of "before-and-after" effects has been retained.

ELIGIBILITY:
Inclusion Criteria:

* people who circulate on French non-motorway non-urban roads during the period of the study
* any person who dies in a road accident on this network during the period of the study, who either dies instantly or within 30 days of the accident, due to the consequences of the accident

Exclusion Criteria:

* all persons involved in an accident on a private road
* all persons involved in a road accident without a motor vehicle

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the population who circulate on French non-motorway non-urban roads during the period of the study may be potentially concerned
Sampling Method: Non-Probability Sample
Enrollment: 80000000 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of the number of fatalities in road accidents before and after the implementation of the measure | before period: 2015-2017 / after period: July 2018- June 2019
  the number of fatalities in road accidents on non-motorway non-urban roads during the period July 2018-June 2019 ("after" the measure) compared to the number of fatalities during the period 2015-2017 ("before" the measure)

SECONDARY OUTCOMES:
Sub-groups analysis of road fatalities, by type of road users, before and after the implementation of the measure | before period: 2015-2017 / after period: July 2018- June 2019
  For each type of road users, the number of fatalities in road accidents on non-motorway non-urban roads during the period July 2018-June 2019 ("after" the measure) compared to the number of fatalities during the period 2015-2017 ("before" the measure)

CONTACTS AND LOCATIONS:
Overall Officials: Marine Millot, PhD, Study Director — Centre d'études et d'expertise sur les risques, l'environnement, la mobilité et l'aménagement
Locations (1):
- Cerema, Lyon, France